CLINICAL TRIAL: NCT00644774
Title: A Comparative, Multi-Center, Pediatric Taste Test Study of Omnicef Versus Zithromax Antibiotic Suspension Medications
Brief Title: A Pediatric Taste Test Study of Omnicef Versus Zithromax Antibiotic Suspension Medications
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Angela M Nilius, Abbott
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: M02-568
Record Dates: First submitted 2008-03-22; First posted 2008-03-27 (Estimated); Last update posted 2008-03-27 (Estimated); Status verified 2008-03

CONDITIONS: Healthy
Keywords: pediatric taste test; antibiotic taste test; cefdinir; azithromycin
MeSH Terms: interventions — Cefdinir; Azithromycin

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: cefdinir (Omnicef)
- 2 (Active Comparator)
  Interventions: Drug: azithromycin

INTERVENTIONS:
Drug: cefdinir (Omnicef) — 2.5 ml of strawberry cream flavored oral suspension 125 mg/5 ml
  Other Names: ABT-198; Omnicef; cefdinir
  Arms: 1
Drug: azithromycin — 2.5 ml of cherry flavored oral suspension 100 mg/5 ml
  Other Names: Zithromax
  Arms: 2

SUMMARY:
To compare the taste and smell acceptability of cefdinir (Omnicef) antibiotic suspension and azithromycin (Zithromax) antibiotic suspension following a single dose of each medication.

DETAILED DESCRIPTION:
The Primary Purpose for the study is "Other". Per ClinicalTrias.gov, more information regarding the primary purpose is described here; this study is a pediatric taste test.

ELIGIBILITY:
Inclusion Criteria:

* Female or male child age 4 through 8 years in good general health.
* Minimum weight of 16.3 kg (36 lb).
* Willing to comply with appropriate instructions provided to complete the study.
* Written informed consent from parent/legal guardian.

Exclusion Criteria:

* Current medical condition, that in the opinion of the Investigator or designee, may interfere with the ability to discriminate taste (e.g., common cold, sinus infection, bronchial infection, etc.).
* History of allergic reaction to cefdinir, azithromycin, prescription (e.g. penicillins or cephalosporins) and/or OTC medications, and/or food products.
* History of significant medical condition (e.g., GI disorders, hematological or bleeding disorders, renal or hepatic diseases).
* Use of any oral medication, vitamins or herbal supplements within 6 hours prior to tasting.
* Temperature > than 99.2°F. Participation in a clinical or marketing research study within the past 3 months.
* Sibling of another subject on the study, or living in the same household as another subject that has participated in a clinical or marketing research study within the past 3 months.
* Family member or close friend employed by an advertising agency, market research company, and/or a company that processes or manufacturers medical or health care products.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 157 (Actual)
Dates: Start 2003-01; Primary Completion 2003-01 (Actual)

PRIMARY OUTCOMES:
Taste and smell acceptance and preference | 2 hours

SECONDARY OUTCOMES:
Adverse events assessment | 72 hours with follow-up to a satisfactory conclusion
Concomitant Medications | 72 hours
Vital signs | 2 hours
Any clinically abnormal observations | 2 hours with follow-up to a satisfactory conclusion

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Scottsdale, Arizona
  - St. Petersburg, Florida
  - Miamiville, Ohio